CLINICAL TRIAL: NCT01843166
Title: Use of Vaginal Estrogen With Pessary Treatment of Pelvic Organ Prolapse and Urinary Incontinence
Brief Title: Vaginal Estrogen With Pessary Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Academic Medical Organization of Southwestern Ontario (Other); University of Western Ontario, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 102186; 18798 (Other: HSREB)
Record Dates: First submitted 2012-07-08; First posted 2013-04-30 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Vaginal Infection; Urinary Tract Infection; Quality of Life
Keywords: Pessary; Patient Satisfaction; Estrogen Cream
MeSH Terms: conditions — Vaginitis; Urinary Tract Infections; Patient Satisfaction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Active Comparator): These patients will utilize a pessary and be given instructions for use and prescription for Premarin vaginal cream 2g at bedtime twice weekly.
  Interventions: Drug: Premarin vaginal cream
- Control group (Placebo Comparator): These patients will utilize a pessary with an inactive placebo cream.
  Interventions: Drug: Placebo cream

INTERVENTIONS:
Drug: Premarin vaginal cream — 2g at bedtime twice weekly
  Arms: Treatment group
Drug: Placebo cream — 2g at bedtime twice weekly
  Arms: Control group

SUMMARY:
Patients presenting with pelvic organ prolapse will be offered the use of a pessary. Vaginal estrogen cream treatment with the pessary will be randomized amongst the patients and patient satisfaction and complication rates will be assessed during follow-up.

DETAILED DESCRIPTION:
This will be a double-blinded, placebo-controlled, randomized controlled trial. Eligible patients presenting to the urogynaecology clinic with pelvic organ prolapse will be offered management with a pessary and participation in the study

Patients who agree to participate in the study will be given a consent form

Patients in the study and thus those who have opted for pessary use will be randomized between two groups:

1. Treatment group - will be given instructions for use and prescription for Premarin vaginal cream 2g at bedtime twice weekly
2. Control group - will utilize pessary with an inactive placebo cream

Both the patient and the investigators will be blinded to patient treatment.

If a patient has expressed willingness to participate in the study over the phone, the research assistant will issue a study number to the patient and pick up the corresponding cream from the LHSC pharmacy to give to the patient at their next clinic visit. The cream will be provided to the patient once they have read the letter of information and signed the consent form.

For follow-up visits, the research assistant will monitor appointment bookings to ensure that the cream is ready in the clinic when the patient has their next follow-up visit.

Patients of both groups will be fitted with a pessary. Pessary fitting will be individualized due to differences in pelvic size and shape and degree of prolapse. Patients may return to the clinic for subsequent fittings until a successful fit has been achieved. An unsuccessful fitting is defined as discontinued pessary use due to discomfort or expulsion.

Patients will be assessed for satisfaction and complications 6 wks, 18 wks, 36 wks and 60 wks after the successful fitting.

To determine patient satisfaction and complications, patients will complete a compilation of validated questionnaires assessing urinary symptoms, sexual function and quality of life at each follow-up.

At each follow-up, a vaginal exam will be done and a vaginal swab and urine sample (for urinalysis and culture and sensitivities) will be taken to assess vaginal bleeding and infections.

ELIGIBILITY:
Inclusion Criteria:

* Any patient presenting to the clinic with pelvic organ prolapse will be offered management with a pessary and will be offered participation in the study.

Exclusion Criteria:

* have a contraindication to the use of estrogen cream or products
* have any allergy to the use of estrogen cream or products
* have a past medical or family history of breast cancer
* have a past medical history of thromboembolism, myocardial infarction and stroke or are pregnant
* have previously used Premarin vaginal cream
* are currently using oral estrogen
* are not competent to consent

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Vaginal infections | 60 weeks
  Vaginal swabs at each follow up visit will be used to detect presence or absence of vaginal infection. A total count of vaginal infections per patient will be compared between groups.

SECONDARY OUTCOMES:
Frequency of urinary tract infection | 60 weeks
  Urine samples at each follow-up visit will be used to detect the presence or absence of a urinary tract infection.
Quality of life | 60 weeks
  Patients will complete validated questionnaires to assess quality of life with respect to urinary, bowel, and sexual function.

CONTACTS AND LOCATIONS:
Overall Officials: Queena Chou, MD, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, University of Western Ontario, London, Ontario, Canada

REFERENCES:
- [Derived] Bugge C, Adams EJ, Gopinath D, Stewart F, Dembinsky M, Sobiesuo P, Kearney R. Pessaries (mechanical devices) for managing pelvic organ prolapse in women. Cochrane Database Syst Rev. 2020 Nov 18;11(11):CD004010. doi: 10.1002/14651858.CD004010.pub4. PMID 33207004